CLINICAL TRIAL: NCT05298514
Title: Investigating Service User Opinions on Sharing Levels of Personal Information
Brief Title: Data Sharing Project Part 2
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: LRS/DP-21/22-26411; 310873 (Other: IRAS)
Record Dates: First submitted 2022-03-08; First posted 2022-03-28 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Data Sharing; Information Dissemination; Mental Health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Not applicable - qualitative research study — We are not delivering interventions. This is a qualitative study in the form of focus groups.

SUMMARY:
Patient data from clinical records are increasingly recognised as a valuable resource and a number of global initiatives exist to promote and enable the sharing of data. However, some mental health service-users have expressed concerns about the use of their data by services, but these have not been explored in depth and the acceptable limits of data sharing remain unclear. The purpose of the study is to present different approaches to data sharing, with examples taken from across the world, varying in levels of anonymity and amounts of data stored and shared, with a view to extracting relevant principles directly from mental health service users. The primary objective of this study is to understand from service-users the limits of acceptable pseudonymised data sharing and data collection methods. This will inform the wider scientific community about any emerging questions and issues on pseudonymised clinical data sharing. We aim to explore the level of benefit service-users would accept, in exchange for the level of pseudonymised data they provide. Additionally, this study aims to investigate what service-users consider "identifiable" data, for example whether they consider demographic or location data or purely their real name to be identifiable. This study will ensure service-user views are an integral contribution to future pseudonymised data sharing systems, maximising applicability and acceptability. This study will use qualitative methods, in the form of focus groups, to gather service-user views. Focus groups will consider what participants believe to be identifiable data, who should get access, how should individuals and/or companies get access, how should data be protected and whether these answers change if pertaining to mental health information. Focus group data will be analysed using thematic analysis. Themes produced will be presented to participants in a second focus group. Participants will be encouraged to expand or change anything.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who have experience of using mental health services or experienced mental health difficulties in the past.
* Aged 18 and above.
* Able to give informed consent.
* Ability to speak fluent English.

Exclusion Criteria:

* If identified through C4C, participants whose care team specify concerns regarding taking part in the study.
* People in whom significant concerns have been raised relating to risk, where risk refers to the extent to which an individual poses a threat to themselves (e.g. self-harm or suicidal intent).
* Inability to give informed consent, as judged by the clinician responsible for a service user's ongoing care, where applicable.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: We want to capture the views of a broad range of service users who have used mental health services or have experienced mental health problems from diverse backgrounds (ethnicity, age and clinical diagnoses).
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Mental health service user opinions on clinical data sharing as explored through qualitative focus groups questions | Through study completion, an average of 1 year
  To understand the requirements of service users, on issues such as privacy, usability, and acceptability of different tiers of data sharing. Furthermore, to investigate what service-users consider "identifiable" data, for example whether they consider identifiable data to be demographic information, location data (consisting of relative and absolute data) or purely their real name.
  This will be achieved by conducting a focus group in which the participants will be asked about hypothetical models of data sharing and their opinions on it. This will be guided by a topic guide asking the following questions:
  1. What is data? What would you consider to be personally identifiable information?
  2. Who gets access?
  3. How should individuals and/or companies get access?
  4. How should data be protected? The focus group will be audio-recorded, transcribed and analysed (via thematic analysis) to answer the primary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Til Wykes, Clinical Doc, Principal Investigator — King's College London